CLINICAL TRIAL: NCT02828527
Title: Care Courses for Mild Head Injury Patients
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Parcours TC léger
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Mild Head Injury
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational

SUMMARY:
Background / Rationale at. The mild head injury.

In France, the incidence of head injuries is estimated at 100,000 per year in France. 80% of mild head trauma. This is a pattern of frequent use of the health system. The reason for consultation, benign appearance, present a significant risk of complication. In 15 to 25% of the evolution of head injury is unfavorable. Disorders of attention, memory disorders, psychiatric events and mood changes may occur. These symptoms are grouped into a syndrome, post-concussion syndrome.

The post-concussion syndrome:

It affects approximately 20,000 people per year in France. This is a common disease and most undervalued in the general population. diagnostic criteria post-concussional disorder according to DSM-IV (Diagnostic and Statistical Manual). Symptoms may persist for more than 3 months after head injury. This syndrome is responsible for suffering, personal and professional sound and quality of life of patients. It is particularly debilitating in everyday life, and can have disastrous consequences on their family, social, cultural and professional. It gives rise to many financial implications with compensation requirements and expertise consultations.

Intention of work In a recent study by a team of neuropsychologists Kremlin Bicetre, it has been shown that screening and early treatment of post-concussion syndrome from the slight head injury prevents chronicity of symptoms.

DETAILED DESCRIPTION:
Methodology :

Design: Cohort study single-center prospective observational. Recruitment period: 15/11/2014 to 15/12/2014 approximately (50 records necessary).

Then follow a month is required. Either theoretical study end: 01/15/2015.

Acquisition of data:

Pre inclusion of patients in the study by sorting CAE emergency department on the following host pattern: traumatic brain injury with loss of consciousness, traumatic brain injury without loss of consciousness, with loss of consciousness discomfort, discomfort without a loss of consciousness peripheral vascular accident PVA.

Collection address, telephone number and an e-mail address of the patient (after delivery of a newsletter).

call the patient and questionnaire submitted between 0 and J15 and J15 and J30 between.

ELIGIBILITY:
Before Inclusion Criteria:

* Traumatic brain injury
* Head injury with loss of consciousness
* Cranio facial trauma
* Peripheral vascular accident
* Discomfort
* Discomfort with loss of consciousness

Before Inclusion Criteria:

* Head trauma notion AND at least one of the following criteria:
* Loss of consciousness <30 minutes
* Glasgow between 13 and 15
* Post Traumatic Amnesia <24H
* Altered mental status at the time of the accident (dizziness, confusion, disorientation)
* Transient focal neurological deficit

Exclusion Criteria:

* <18
* Major Trust
* Context of acute alcohol (> 3 glasses) or toxic taking (drugs)
* Not understanding or communication
* Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to emergency Unit of Hopital Paris Saint Jospeh
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-09-12 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of change in Glasgow score | submitted between Day 0 and Day 15 and between Day 15 and Day 30

CONTACTS AND LOCATIONS:
Overall Officials: AÏM Jean luc, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France